Title: Efficacy and Safety of Nadroparin Calcium-Warfarin Sequential

Anticoagulation in Portal Vein Thrombosis in Cirrhotic Patients: A

Randomized Controlled Trial

NCT number: NCT04173429

Date of the Document:2020-7-3

## Statistical Analysis Plan

Statistical analysis was performed using the statistical software IBM SPSS Statistical 24.0. The analysis of the outcomes between NWS therapy group and control group was conducted by both intention-to-treat (ITT) and per-protocol (PP) analysis. All eligible patients were analyzed by ITT analysis, and patients who did not violate the protocol were analyzed by PP analysis.

Quantitative variables were expressed as the mean  $\pm$  standard deviation (SD), while qualitative variables were expressed as percentages. Quantitative variables were compared using Student's t-test or Wilcoxon-rank sums test, and categorical variables were compared using chi-squares or Fisher's exact test, as appropriate. Univariate and multivariate logistic regression analysis were performed to find significant end point predictors for recanalization. A two-tailed p-value <0.05 was considered statistically significant.